CLINICAL TRIAL: NCT04610060
Title: Effectiveness of Standardized Outpatient Cardiac Rehabilitation Program Combined With Power Walking on Quality of Life and Exercise Capacity in Patients With Post-coronary Angioplasty: A Pragmatic Randomized Controlled Trial
Brief Title: Power Walking in Cardiac Patients Who Underwent Post-coronary Angioplasty
Acronym: PowerWalk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INT/COHS/PG/015-2020
Record Dates: First submitted 2020-09-25; First posted 2020-10-30 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Heart Diseases, Ischemic; Coronary Artery Disease; Coronary Arteriosclerosis; Coronary Syndrome; Coronary Disease
Keywords: cardiac rehabilitation; coronary angioplasty; power walking; heart quality of life; metabolic equivalents task
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Angina, Unstable; Coronary Disease

STUDY DESIGN:
Intervention Model Description: A 4-Week, Single-Blind, Parallel-Group Study
Who Masked: Participant, Investigator
Masking Description: For each participant were blinded till allocation of treatment. Investigator was also blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power walking group (Experimental): Exercise in the form of Power walking at hospital for 10-20 minutes on treadmill with various exercise intensities. Weekly Steps at home 30 minutes walking with target to reach 1000 steps daily.
  Standardised Outpatient Cardiac Rehabilitation based on ACSM Guidelines where provided for four weeks. The program consisted of warm up, aerobics, strengthening and cool down exercises based on ACSM Guidelines described in Table 1 (Deborah, Jonathan, Gary & Meir, 2018).
  Interventions: Behavioral: Power walking; Behavioral: Standardised outpatient cardiac rehabilitation
- Standardised outpatient cardiac rehabilitation group (Active Comparator): Standardised Outpatient Cardiac Rehabilitation based on ACSM Guidelines where provided for four weeks. The program consisted of warm up, aerobics, strengthening and cool down exercises based on ACSM Guidelines described in Table 1 (Deborah, Jonathan, Gary & Meir, 2018).
  Interventions: Behavioral: Standardised outpatient cardiac rehabilitation

INTERVENTIONS:
Behavioral: Power walking — Exercise in the form of Power walking at hospital for 10-20 minutes on treadmill with various exercise intensities. Weekly Steps at home 30 minutes walking with target to reach 1000 steps daily.
  It is a form of exercise where active upper body movement is performed along with usual walking. It is a fast walking exercise done at a speed of 6 to 8 km/h. During power walking the back is kept straight with the centre of gravity moving from heal, sole, and to hallux. There is active swing back and forth movement of elbow joint with 90 degrees of flexion while walking.
  Weekly protocol for power walking
  * Week 1 60-65 % of the target heart rate (THR) 5,000 to 7,499 steps/day
  * Week 2 65-70 % of the target heart rate (THR) 7,500 to 9,999 steps/day
  * Week 3 70-75 % of the target heart rate (THR) >=10,000 steps/day
  * Week 4 75-80 % of the target heart rate (THR) >12,500 steps per day
  Arms: Power walking group
Behavioral: Standardised outpatient cardiac rehabilitation — Standardised Outpatient Cardiac Rehabilitation based on ACSM Guidelines the intervention group received the following four weeks of intense training program

SUMMARY:
The risk and prevalence of cardiovascular disease in United Arab Emirates (UAE) is high with ischemic heart disease ranks first in terms of major cause of mortality. Large number of patients undergoes coronary angioplasty but very few participate in cardiac rehabilitation because its awareness is not widespread in middle east region.

The objectives was to find the influence of standardized outpatient cardiac rehabilitation program along with power walking on Heart quality of life (Heart QoL), functional exercise capacity, Left Ventricular Ejection Fraction and metabolic equivalent task (MET's) among patients with post coronary angioplasty.

The investigators conducted a randomized clinical trail in out patient physiotherapy department at Thumbay hospitals Dubai, on patients who underwent coronary artery angioplasty. After meeting the inclusion criteria, participants were randomized into standardized outpatient cardiac rehabilitation program along with power walking (intervention group) or standardized outpatient cardiac rehabilitation program (control group).

A 4 weeks of 12 outpatient cardiac rehabilitation sessions consisting of 3 sessions per week was provided to both the groups. Intervention group received standardized outpatient cardiac rehabilitation program along with power walking based on targeted heart rate and weekly steps, whereas control group received only standardized outpatient cardiac rehabilitation program based on American College of Sports Medicine (ACSM) Guidelines.

The investigators measured Quality Of Life (HRQoL) by HeartQoL questionnaire, Exercise Capacity by 6 min walk test (6MWT), Left ventricle Ejection fraction (LVEF) using Echocardiogram, Metabolic Equivalent Task (MET'S) using Symptom-limited exercise stress test and Average number of steps walked daily using step up smartphone Pedometer App.

DETAILED DESCRIPTION:
Approximately 17.8 million worldwide deaths per year are due to cardiovascular disease (CVD). Arab countries are at higher risk of CVD in which middle income countries are mostly at burden. "The threshold for cardiac arrests and cardiovascular disease (CVD) worldwide is 65 years, while people in the UAE are suffering from the CVD at the age of 45" reported by Emirates Cardiac Society. One of the most common causes of cardiovascular deaths is coronary artery disease (CAD). Coronary angioplasty one of the most common non-surgical approach for the treatment of ischemic coronary artery disease. It is widely accepted that cardiac rehabilitation can be beneficial for patients with heart diseases. Most of the patients won't achieve adequate functional improvement, if rehabilitation exercises are not done on regular basis post-coronary angioplasty.

In cardiac rehabilitation (CR) programs, psychosocial function and the assessment of quality of life (QOL) are the major objective parameters commonly used by researchers. Physical activity and emotional status influence health related quality of life (HRQOL) in patient underwent coronary angioplasty. It is important to find effectiveness of CR on health related quality of life (HRQOL). Studies has shown that tailored exercise training helped to improve Left Ventricle Ejection Fraction (LVEF) in patients post coronary angioplasty. A systematic review highlighted the effectiveness of using 6MWT to show improvement of functional capacity in patients undergoing cardiac rehabilitation.

It is well known that walking exercise reduces cardiovascular disease-related mortality and predicts longevity in patients with established CAD. One of the integral components of cardiac rehabilitation is treadmill walking. A meta-analysis demonstrated that physical activity could be enhanced in patients with the use of pedometer. Recent evidence shows that smartphone apps are effective at promoting physical activity. Studies also shows that smartphone Apps are more accurate in tracking steps as compared to fitness trackers.

Power walking is an effective part of phase II cardiac rehabilitation. Running is preferred over walking since oxygen consumption while running is less as compared to walking.

It was reported that up to 1 year, cardiac rehabilitation improves QOL in patients with acute myocardial infarction (AMI) or revascularization procedures. Four weeks of short CR course provides better attendance, improvement in quality of life and exercise capacity.

Accordingly, the current study was conducted for 4 weeks, a shorter period of rehabilitation and documented the effectiveness on cardiac fitness including health related quality of life, functional exercise capacity, ejection fraction and metabolic equivalent task (MET's) of patients with post angioplasty.

Although the advantages of CR are well known to most of the physicians, still one third of the patients do not receive CR post coronary angioplasty due to poor referral trends. Higher rates of quality-of-care measures were found among patients who were referred for CR compared to those who were not referred. Post coronary angioplasty patients need to continue with cardiac rehabilitation in a progressive manner to attain the overall improvement. In a comparative study where 5 and 39 CR programs participated from Arab countries and Canada respectively showed that in Arab countries CR programs are very limited. Recent statistics in UAE has shown that 30% deaths are due to cardiovascular diseases, 30-70% population has cardiovascular diseases or are at risk and 37% population do not exercise and are physical inactive.

The concept is very clear that significant number of eligible patients with cardiac conditions is not referred for outpatient CR. Although most patients post coronary angioplasty are encouraged by cardiologist to gradually increase their activity levels, limited data are available on the amount of physical and walking activity and regular aerobic exercises done by patients with post coronary angioplasty at phase II CR.

Power walking has an advantage that it consumes 55% more energy in comparison to just walking alone or running at a speed of 6 to 8 km/h, while being at a lower intensity. Despite the advantages of power walking, the exercise effects have not been reported in cardiac rehabilitation programs.

This study will help to fulfill great need for referral and awareness of out patient cardiac rehabilitation by proving outcomes of standardized outpatient cardiac rehabilitation program. The investigators utilized power walking along with standardized cardiac rehabilitation to find effectiveness on health related quality of life, functional exercise capacity, ejection fraction and metabolic equivalent task (MET's) of patients with post coronary angioplasty. Henceforth, the need for research is to prove the effectiveness of cardiac rehabilitation in UAE population.

ELIGIBILITY:
Inclusion Criteria:

* Those patients underwent coronary angioplasty and willing to participate
* Age between 18-70 years.
* Both the genders.
* Patients who completed not < 2 week and not >12 weeks post hospital discharge.
* Patients not limited to diabetes mellitus, controlled Hypertension, Hyperlipidemia and obese.
* Availability of smart phone.

Exclusion Criteria:

* Malignancy.
* Neurological disorders.
* Psychoneurotic disorders Causing deficit in functioning.
* Significant valvular diseases.
* Active pericarditis or myocarditis.
* Patient with complications related to angioplasty procedure.
* Severe orthostatic hypotension.
* Severe obstructive airway disease or any other chronic pulmonary disorder.
* Physically disabled patients.
* All Musculoskeletal disorders affecting movement of bilateral upper and lower limbs while walking at a faster speed of 6 to 8 km/h (47)
* Patients contraindicated for exercises testing and training.
* Severe uncontrolled hypertension (Systolic Blood Pressure >180 mmHg and/or Diastolic Blood Pressure >100 mmHg).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-13 (Actual)

PRIMARY OUTCOMES:
Heart Quality of Life questionnaire global scores | From the start of treatment i.e., Day 1, Base line assessment until 4th week, i.e., completion of 12th therapy session
  HeartQoL questionnaire has 14-items with two subscales consisting of 10 and 4 -item of physical and emotional subscales respectively. Subscale scores are summarised to global scores. Standard deviation scores specific to population mean were used for statistical analysis.

SECONDARY OUTCOMES:
Six Minute Walk Test (6MWT) distance in meters | From the start of treatment i.e., Day 1, Base line assessment until 4th week, i.e., completion of 12th therapy session
  The outcome of the 6MWT is the 6-minute walk distance (6MWD) measured in meters.
Percentage of Left ventricle Ejection fraction (LVEF) i.e., Percentage of blood pumped out of left ventricle during each contraction. | From the start of treatment i.e., Day 1, Base line assessment until 4th week, i.e., completion of 12th therapy session
  Percentage of blood pumped out of left ventricle during each contraction measured by echocardiogram.
Walking steps per day measured by pedometer | From the start of treatment i.e., Day 1, Base line assessment until 4th week, i.e., completion of 12th therapy session
  A digital mobile application was used to record steps taken on day by day basis and cumulative average until 4th week was calculated
Energy expenditure measured in Metabolic equivalent of task (MET) | From the start of treatment i.e., Day 1, Base line assessment until 4th week, i.e., completion of 12th therapy session
  MET was calculated based on symptom-limited exercise stress test, i.e, Bruce protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Kumaraguruparan Gopal, Ph.D, Principal Investigator — Gulf Medical University; Ramprasad M, Ph.D, Study Director — Gulf Medical University
Locations (1):
- Gulf Medical University, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Physiotherapy research international, issue 26(4), e1919, 2021 — https://pubmed.ncbi.nlm.nih.gov/34231290/